CLINICAL TRIAL: NCT04366284
Title: Optimizing the Scalability of Evidence-Based Behavioral Sleep Medicine Practices With a Digital Health Platform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Noctem, LLC (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Naval Health Research Center (U.S. Federal Agency); US Air Force Medical Readiness Agency (Unknown); KNOWESIS, Inc. (Unknown)
Responsible Party: Principal Investigator, Anne Germain, Principal Investigator, Noctem, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-406; MT190002.01 (Other Grant/Funding Number: MTEC/MOMRP)
Record Dates: First submitted 2020-04-15; First posted 2020-04-28 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-06

CONDITIONS: Implementation; Digital Health; Chronic Insomnia
Keywords: Cognitive-Behavioral Therapy for Insomnia; Implementation-Effectiveness; Dissemination and Implementation Research
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NOCTEM only (NOCTEM) (Active Comparator): No external or internal facilitation
  Interventions: Other: No Facilitation Support
- External Facilitation (NOCTEM+EF) (Active Comparator): External facilitation only
  Interventions: Other: External Facilitation Support
- External and Internal Facilitation (NOCTEM+EF/IF) (Active Comparator): External and internal facilitation
  Interventions: Other: External and Internal Facilitation Support

INTERVENTIONS:
Other: No Facilitation Support — Clinicians will have full use of the NOCTEM platform. They will not have scheduled and/or structured contacts with the facilitation teams, however can reach out to the NOCTEM team or their local point of contact and coordinator with questions or technical issues that may arise.
  Arms: NOCTEM only (NOCTEM)
Other: External Facilitation Support — Clinicians will have full use of the NOCTEM platform and the NOCTEM team will provide external facilitation via bi-weekly consult or supervision teleconference, or via telephone. The NOCTEM team will also be available by email and text messaging on an as needed basis.
  Arms: External Facilitation (NOCTEM+EF)
Other: External and Internal Facilitation Support — Clinicians will have full use of the NOCTEM platform and external facilitation support. In addition to external facilitation by the NOCTEM team a local point of contact and coordinator will serve as a more proximal facilitator.
  Arms: External and Internal Facilitation (NOCTEM+EF/IF)

SUMMARY:
The purpose of this study is to compare three different ways to deploy a clinician-decision support platform called NOCTEM COAST among behavioral health care providers who encounter patients with insomnia.

DETAILED DESCRIPTION:
Insomnia and other sleep disorders are highly prevalent among military service members and compromise readiness, health, and performance; increase the risk of injury; and are associated with astronomical healthcare costs. The first-line treatment recommended for insomnia is cognitive-behavioral treatment for insomnia (CBTI). However, the large number of service members who are in need of this treatment outnumber the clinicians who are experts in behavioral sleep medicine and who currently provide this intervention in a cost-efficient manner and in a way that is acceptable and accessible to patients and clinicians. To address this challenge and scale the delivery and access to evidence-based behavioral sleep interventions, NOCTEM™ has developed a digital health platform called COAST (Clinician Operated Assistive Sleep Technology). However, the most effective way to implement the use of digital sleep health technology, and its comparative impact on patient outcomes, remain to be determined. Therefore, this trial will compare three different ways to deploy the NOCTEM™ platform among behavioral health care providers who encounter patients with insomnia. Specifically, the study will evaluate and compare without external or internal support (NOCTEM), with external support (i.e., facilitation) offered by the NOCTEM team (NOCTEM+EF), and with external support and internal support from local champions (NOCTEM+EF/IF). The trial will also compare the overall magnitude of improvements in insomnia among patients who use the NOCTEM app with their provider.

ELIGIBILITY:
Inclusion Criteria:

For clinicians:

* Completion of the first half of the workshop or similar Behavioral Sleep Medicine workshop in the past 6 months
* Completion of the second half of the workshop, including a training session to learn about the use of the NOCTEM platform
* See patients who present with insomnia
* Use cognitive-behavioral techniques as part of their practice

For patients:

* Are service members, veterans, or adult dependents who receive behavioral health care at one of the participating sites
* Present with complaints of insomnia
* Own a smart phone or smart device
* Deemed suitable by their clinician to receive the sleep intervention via the NOCTEM platform
* Confirm their willingness to use the NOCTEM app for sleep care with their provider

Exclusion Criteria:

For clinicians:

* Do not provide direct behavioral health care to service members
* Do not complete the two-part workshop and the 2-week proficiency training

For patients (recommended):

* Suspected, diagnosed, or inadequately untreated sleep apnea (less than 4 hours of continuous positive airway pressure [CPAP] use per night)
* Psychotic symptoms
* A history of bipolar disorders
* Women who are pregnant or breastfeeding and parents of children younger than 3 months of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach among clinicians randomized to NOCTEM only, NOCTEM+EF, or NOCTEM+EF/IF | 3 month follow-up
  The ratio of clinicians who consent to participate and complete the NOCTEM training over the number of clinicians who received information about the training.
Adoption among clinicians randomized to NOCTEM only, NOCTEM+EF, or NOCTEM+EF/IF | 3 month follow-up
  The ratio of newly trained clinicians who use the NOCTEM system over the total number of clinicians who completed the NOCTEM training.
Maintenance (sustainability) among clinicians randomized to NOCTEM only, NOCTEM+EF, or NOCTEM+EF/IF | 6-month follow-up
  Comparison of frequency of use of the NOCTEM platform by the trained clinicians, across the three groups (NOCTEM vs. NOCTEM+EF vs. NOCTEM+EF/IF).
Change in Insomnia Severity Index | From Baseline to Post-Acute Intervention at Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Health Research Center, San Diego, California, United States

REFERENCES:
- [Derived] Germain A, Markwald RR, King E, Bramoweth AD, Wolfson M, Seda G, Han T, Miggantz E, O'Reilly B, Hungerford L, Sitzer T, Mysliwiec V, Hout JJ, Wallace ML. Enhancing behavioral sleep care with digital technology: study protocol for a hybrid type 3 implementation-effectiveness randomized trial. Trials. 2021 Jan 11;22(1):46. doi: 10.1186/s13063-020-04974-z. PMID 33430955